CLINICAL TRIAL: NCT03878602
Title: Delayed Umbilical Cord Clamping in Elective Caesarean Section: What Are the Benefits
Brief Title: Umbilical Cord Clamping: What Are the Benefits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Poliambulanza Istituto Ospedaliero (Other)
Responsible Party: Principal Investigator, Giuseppe De Bernando, Principal Investigator, Fondazione Poliambulanza Istituto Ospedaliero
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3176
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Results first posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Delayed Cord Clamping
Keywords: Newborn; Elective Caesaren Section; Cord Clamping
MeSH Terms: interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Newborns will be subjected to umbilical cord immediate clamping
  Interventions: Procedure: Immediate umbilical cord clamping
- Study Group (Experimental): Newborns will be subjected to umbilical cord delayed clamping
  Interventions: Procedure: Delayed umbilical cord clamping

INTERVENTIONS:
Procedure: Delayed umbilical cord clamping — Umbilical cord will be clamped after 1 min after the birth of the newborn
  Arms: Study Group
Procedure: Immediate umbilical cord clamping — Umbilical cord will be clamped immediately after the birth of the newborn
  Arms: Control Group

SUMMARY:
Umbilical cord clumping consists in the binding of the umbilical cord by nipper to interrupt blood flow from placenta to foetus. Umbilical cord can be clamped within 30s or at least 1 min after birth. A lot of studies have shown that delayed umbilical cord clamping is associated with greater haemoglobin concentration, better iron storage between 3-6 months of life and lower incidence for transfusion and neonatal hypotension compared to immediate umbilical cord clumping. Newborns subjected to Caesarean Section showed greater value of haemoglobin and lower value of red blood cells compared to newborns birth by vaginal delivery. Despite evidence of beneficial effects for delayed umbilical cord clamping after eutocic delivery, this practice is not yet taken into consideration after elective Caesarean Section.

DETAILED DESCRIPTION:
Umbilical cord cutting determines the separation of the newborn from mother. Umbilical cord clumping consists in the binding of the umbilical cord by nipper to interrupt blood flow from placenta to foetus. In the spontaneous labor there are two modalities to obtain umbilical cord clamping: the first modality is immediate umbilical cord clamping within 30s from birth. The second modality is delayed umbilical cord clamping at least 1 min after birth. After 1 min, cerebral blood flow is reduced again because of lower cardiac output.

A lot of studies have shown that delayed umbilical cord clamping is better than the early umbilical clamping because delayed umbilical cord clamping is associated with a great haemoglobin concentration in the newborns and best iron storage between 3-6 months of life and less incidence for transfusion and neonatal hypotension. Experimental studies, executed on animals and humans, analysed cardiocirculatory changes in the foetus immediately after birth and the importance of the delayed clamping for the hemodynamic stabilization, particularly in the lowest gestational age.

In a recent randomized study conducted in Nepal on 540 newborns, birth by eutocic delivery with 39.2 weeks of gestational age, showed that delayed umbilical cord clamping after 3 min of life is correlated with a better haemoglobin level and less incidence of anaemia at 8 months of life. Zhou et al. conducted a meta-analysis that included hematologic parameters obtained by umbilical cord, placenta and newborns blood.

Association of Italian Hospital Gynecologists Obstetricians (AOGOI) declared contraindicated conditions to execute a delayed umbilical cord clamping:

Hypoxic-ischemic events: detachment of placenta, prolapse of the funiculus, uterine rupture, shoulder dystocia, premature rupture of fetal membranes, placenta previa, maternal collapse, embolism amniotic, maternal cardiac arrest. Monochorionic twins, Fetal Hydrops, Umbilical cord damaged, Isoimmunization Rh.

Researchers concluded that newborns subjected to Caesarean Section showed greater value of haemoglobin and lower value of red blood cells compared to newborns birth by vaginal delivery. Haematocrit difference was greater between newborns birth by elective Caesarean Section compared to those birth by Caesarean Section in labor. Nowadays, researchers found no side effects of delayed umbilical cord clamping except a slight increase of phototherapy needs.

Despite evidence of beneficial effects for delayed umbilical cord clamping after eutocic delivery, this practice is not yet taken into consideration after elective Caesarean Section. The aim of the study protocol is to investigate the effects of the clamping after 1 min from birth by elective Caesarean Section on heart rate, saturation, body temperature, bilirubin, haematocrit and glycemia.

ELIGIBILITY:
Inclusion Criteria:

* Birth Body Weight = appropriate for gestational age
* Delivery mode= Elective Caesarean Section
* Mothers' BMI = 19-24,9
* Mothers'age ≤ 37 years

Exclusion Criteria:

* Admission in NICU;
* Neonatal Resuscitation
* Hypoxic-ischemic events: detachment of placenta, prolapse of the funiculus, uterine rupture, shoulder dystocia, premature rupture of foetal membranes, placenta previa, maternal collapse, embolism amniotic, maternal cardiac arrest
* Pathologies ;
* Smoking mothers;
* Assumption of drugs during pregnancy
* Mother toxicomaniac

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 142 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe De Bernardo, M.D., Principal Investigator — Poliambulanza Foundation; Maurizio Giordano, B.Sc., Study Chair — University of Naples Federico II, School of Medicine; Laura Linetti, Dr., Study Director — Poliambulanza Foundation
Locations (1):
- Department of mother and child's Health Poliambulanza Foundation, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Katheria A, Hosono S, El-Naggar W. A new wrinkle: Umbilical cord management (how, when, who). Semin Fetal Neonatal Med. 2018 Oct;23(5):321-326. doi: 10.1016/j.siny.2018.07.003. Epub 2018 Jul 20. PMID 30076109
- [Result] Bhatt S, Alison BJ, Wallace EM, Crossley KJ, Gill AW, Kluckow M, te Pas AB, Morley CJ, Polglase GR, Hooper SB. Delaying cord clamping until ventilation onset improves cardiovascular function at birth in preterm lambs. J Physiol. 2013 Apr 15;591(8):2113-26. doi: 10.1113/jphysiol.2012.250084. Epub 2013 Feb 11. PMID 23401615
- [Result] Polglase GR, Dawson JA, Kluckow M, Gill AW, Davis PG, Te Pas AB, Crossley KJ, McDougall A, Wallace EM, Hooper SB. Ventilation onset prior to umbilical cord clamping (physiological-based cord clamping) improves systemic and cerebral oxygenation in preterm lambs. PLoS One. 2015 Feb 17;10(2):e0117504. doi: 10.1371/journal.pone.0117504. eCollection 2015. PMID 25689406
- [Result] Alzaree F, Elbohoty A, Abdellatif M. Early Versus Delayed Umbilical Cord Clamping on Physiologic Anemia of the Term Newborn Infant. Open Access Maced J Med Sci. 2018 Aug 15;6(8):1399-1404. doi: 10.3889/oamjms.2018.286. eCollection 2018 Aug 20. PMID 30159064
- [Result] Ghavam S, Batra D, Mercer J, Kugelman A, Hosono S, Oh W, Rabe H, Kirpalani H. Effects of placental transfusion in extremely low birthweight infants: meta-analysis of long- and short-term outcomes. Transfusion. 2014 Apr;54(4):1192-8. doi: 10.1111/trf.12469. PMID 24843886
- [Result] Backes CH, Rivera BK, Haque U, Bridge JA, Smith CV, Hutchon DJR, Mercer JS. Placental transfusion strategies in very preterm neonates: a systematic review and meta-analysis. Obstet Gynecol. 2014 Jul;124(1):47-56. doi: 10.1097/AOG.0000000000000324. PMID 24901269
- [Result] Nevill E, Meyer MP. Effect of delayed cord clamping (DCC) on breathing and transition at birth in very preterm infants. Early Hum Dev. 2015 Jul;91(7):407-11. doi: 10.1016/j.earlhumdev.2015.04.013. Epub 2015 May 15. PMID 25984654
- [Result] Wafaa Taha Ibrahim Elgzar, Heba Abdel-Fatah Ibrahim, Hanan Heiba Elkhateeb."Effects of Deferred Versus Early Umbilical Cord Clamping on Maternal and Neonatal Outcomes" - American Journal of Nursing Research, 2017,5(4), 115-128
- [Result] Valero J, Desantes D, Perales-Puchalt A, Rubio J, Diago Almela VJ, Perales A. Effect of delayed umbilical cord clamping on blood gas analysis. Eur J Obstet Gynecol Reprod Biol. 2012 May;162(1):21-3. doi: 10.1016/j.ejogrb.2012.01.020. Epub 2012 Mar 8. PMID 22405491
- [Result] Kc A, Rana N, Malqvist M, Jarawka Ranneberg L, Subedi K, Andersson O. Effects of Delayed Umbilical Cord Clamping vs Early Clamping on Anemia in Infants at 8 and 12 Months: A Randomized Clinical Trial. JAMA Pediatr. 2017 Mar 1;171(3):264-270. doi: 10.1001/jamapediatrics.2016.3971. PMID 28114607
- [Result] Zhou YB, Li HT, Zhu LP, Liu JM. Impact of cesarean section on placental transfusion and iron-related hematological indices in term neonates: a systematic review and meta-analysis. Placenta. 2014 Jan;35(1):1-8. doi: 10.1016/j.placenta.2013.10.011. Epub 2013 Nov 20. PMID 24290868
- [Result] McDonald SJ, Middleton P, Dowswell T, Morris PS. Effect of timing of umbilical cord clamping of term infants on maternal and neonatal outcomes. Cochrane Database Syst Rev. 2013 Jul 11;2013(7):CD004074. doi: 10.1002/14651858.CD004074.pub3. PMID 23843134
- [Derived] De Bernardo G, Giordano M, De Santis R, Castelli P, Sordino D, Trevisanuto D, Buonocore G, Perrone S. A randomized controlled study of immediate versus delayed umbilical cord clamping in infants born by elective caesarean section. Ital J Pediatr. 2020 May 24;46(1):71. doi: 10.1186/s13052-020-00835-2. PMID 32448358

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate Clamping: Newborns will be subjected to umbilical cord immediate clamping
  Immediate umbilical cord clamping: Umbilical cord will be clamped immediately after the birth of the newborn
- Delayed Clamping: Newborns will be subjected to umbilical cord delayed clamping
  Delayed umbilical cord clamping: Umbilical cord will be clamped after 1 min after the birth of the newborn
Period: Overall Study
Arm/Group | Immediate Clamping | Delayed Clamping
Started | 75 | 67
Completed | 66 | 66
Not Completed | 9 | 1
Not completed — cord blood donation | 7 | 1
Not completed — incomplete data collection | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Study Group | Total
Number analyzed (Participants) | 66 | 66 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 66 | 66 | 132
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 30 | 62
  Male | 34 | 36 | 70
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 66 | 66 | 132
Region of Enrollment [Number; unit: participants]
  Italy | 66 | 66 | 132

OUTCOME MEASURES:

1. Primary Outcome: Change of Heart Rate After Delayed Umbilical Clamping
Description: It will be measured the change of heart rate (HR)
Time Frame: 5 minutes and 10 minutes after birth
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 66 | 66
bpm
  5 minutes | 164 (18) | 157 (15)
  10 minutes | 163 (15) | 155 (13)

2. Primary Outcome: Change of Saturation After Delayed Umbilical Clamping
Description: Saturation change (SpO2)
Time Frame: 5 minutes and 10 minutes after birth
Measure: Mean (Standard Deviation); unit: percent of saturated hemoglobin
Arm/Group | Immediate Clamping | Delayed Clamping
Number analyzed (Participants) | 66 | 66
percent of saturated hemoglobin
  5 minutes | 88.98 (7.027) | 89.169 (7.453)
  10 minutes | 95.238 (3.976) | 96.046 (3.346)

3. Primary Outcome: Change of Temperature After Delayed Umbilical Clamping
Description: Temperature change (T)
Time Frame: 5 minutes after birth
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Immediate Clamping | Delayed Clamping
Number analyzed (Participants) | 66 | 66
degrees Celsius | 36.60 (0.64) | 36.64 (0.64)

4. Secondary Outcome: Misuration of the Hemo Gluco Test After Delayed Umbilical Clamping
Description: hemo gluco test (HGT)
Time Frame: 120 minutes after birth
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Immediate Clamping | Delayed Clamping
Number analyzed (Participants) | 66 | 66
mg/dl | 60.32 (9.937) | 56.02 (17.101)

5. Secondary Outcome: Misuration of the Hematocrit After Delayed Umbilical Clamping
Description: hematocrit (Ht)
Time Frame: 72 hours of life
Measure: Mean (Standard Deviation); unit: percent of occupied blood volume
Arm/Group | Immediate Clamping | Delayed Clamping
Number analyzed (Participants) | 66 | 66
percent of occupied blood volume | 51.56 (6.929) | 56.71 (6.663)

6. Secondary Outcome: Misuration of the Bilirubin After Delayed Umbilical Clamping
Description: bilirubin
Time Frame: 72 hours of life
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Immediate Clamping | Delayed Clamping
Number analyzed (Participants) | 66 | 66
mg/dl | 7.06 (2.76) | 8.54 (2.90)

ADVERSE EVENTS:
Time Frame: adverse event data were collected through discharge
Arm/Group | Control Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 0/66 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT03878602/Prot_SAP_000.pdf